CLINICAL TRIAL: NCT04032912
Title: Eliminating the Need for Conventional Histopathological Assessment of Diminutive Colon Polyps - The Non-Optical Resect and Discard Study (NORD)
Brief Title: The Non-Optical Resect and Discard Study (NORD)
Acronym: NORD
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 16.367
Record Dates: First submitted 2019-07-04; First posted 2019-07-25 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2018-04

CONDITIONS: Polyp of Colon
Keywords: Polyp resection; Colorectal cancer
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: iScan — this instrument provides extra confidence for in vivo diagnosis through improved vessel and mucosal pattern characterization.
  Other Names: Optivista

SUMMARY:
Eliminating the need for conventional histopathological assessment of diminutive colon polyps - The Non-Optical Resect and Discard (NORD) study

DETAILED DESCRIPTION:
Implementation of this approach by community-based gastroenterologists has failed to reach the required quality benchmarks and studies evaluating optical biopsy have not shown diagnostic test performance results that meet standards set by society guidelines in order to promote its widespread clinical adoption. Optical polyp diagnosis and the current resect and discard approach are too complex for clinical adoption. Thus, clinical implementation of this valuable concept has not been achieved to date and its cost-saving potential has not been realized. In order to effectively operationalize a resect and discard strategy, one must find a different way to distinguish neoplastic from non-neoplastic polyps. There exist differences in the proportion of polyps found to be adenomatous in the left and right colon. One recent study reported that 30% of left-sided polyps and 76% of right-sided polyps were found to be adenomas on histology. Since polyps located in the proximal colon are more likely to be adenomas and polyps in the recto-sigmoid colon are more likely hyperplastic we hypothesized that a model based on polyp location might be able to replace optical biopsy and histopathology. Such an approach would be very simple to adopt by every clinician and would allow for easy adoption into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age 45 to 80 years
* Indication for full colonoscopy

Exclusion Criteria:

* Known inflammatory bowel disease
* Active colitis
* Coagulopathy
* Familial polyposis syndrome
* Poor general health defined as an ASA class > 3
* Emergency colonoscopies.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 45-80 year old patients scheduled for an elective colonoscopy with the potential of a polyp removal will be considered for the study. This includes patients hospitalized that do not require an emergency colonoscopy (defined as colonoscopy in the emergency or intensive care unit or patients with active upper or lower gastrointestinal bleeding). Potential study subjects are approached to participate: 1) during an outpatient clinic; 2) at their arrival at the endoscopy clinic on the day of the colonoscopy; or 3) on the hospital ward (for patients hospitalized).
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Examine concordance with the pathology-based surveillance recommendation of two new resect and discard models | 24 months
  Our aim is to examine and to make a comparison of these models with the currently endorsed resect and discard approach that is based on optical polyp diagnosis and we will also obtain histopathology for all polyps as a reference gold-standard to which all models are compared.

SECONDARY OUTCOMES:
Assess for how many patients each model will theoretically reduce the need for histopathologic assessment and follow-up consultations to discuss pathology results and surveillance interval recommendations | 24 months
  Assess for how many patients each model will theoretically reduce the need for histopathologic assessment and follow-up consultations to discuss pathology results and surveillance interval recommendations
Re-evaluate classical optical biopsy criteria (NICE and SANO classifications) | 24 months
  We will assess this in conjunction with different digital chromoendoscopy methods (NBI, iScan and Optivista) and assess concordance between these imaging methods and classification systems to differentiate neoplastic from non-neoplastic polyps.
Assess which factors are associated with accuracy and negative predictive value (NPV) of optical polyp diagnosis | 24 months
  Assess which factors are associated with accuracy and negative predictive value (NPV) of optical polyp diagnosis
Evaluate Polyp-Based Resect and Discard model | 24 months
  Surveillance interval agreement of the PBRD strategy compared with pathology-based management according to the 2020 USMSTF guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Taghiakbari M, Pohl H, Djinbachian R, Barkun A, Marques P, Bouin M, Deslandres E, Panzini B, Bouchard S, Weber A, von Renteln D. The location-based resect and discard strategy for diminutive colorectal polyps: a prospective clinical study. Endoscopy. 2022 Apr;54(4):354-363. doi: 10.1055/a-1546-9169. Epub 2021 Aug 26. PMID 34448185